CLINICAL TRIAL: NCT03195426
Title: Is There a Real Diaphragm-Sparing Nerve Block for Arthroscopic Shoulder Surgery?
Brief Title: A Diaphragm-Sparing Nerve Block for Arthroscopic Shoulder Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Medipole Garonne (Other)
Responsible Party: Principal Investigator, Dr Marty Philippe, Dr Marty Philippe, Clinique Medipole Garonne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-202
Record Dates: First submitted 2017-06-15; First posted 2017-06-22 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Intervention Model Description: This study aims at assessing the effectiveness of combined SSNB, ICB and supraclavicular nerve block (SCNB) as surgical anesthesia for patients scheduled for arthroscopic shoulder surgery. The secondary objective was to test the hypothesis that SSNB-ICB-SCNB combination could spare phrenic nerve.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- distal nerves blocks group (Experimental): This study aims at assessing the effectiveness of combined supra scapular nerve block, infraclavicular block and supraclavicular nerve block as surgical anesthesia for patients scheduled for arthroscopic shoulder surgery.
  These blocks are performed for decades in routine care. The originality of this study is to analyze the combination of these different blocks for post-operative pain relief in arthroscopic shoulder surgery. This combination can be considered as an alternative to interscalene block well known to be associated with diaphragmatic paralysis.
  Local anesthetics used in this study are used for many years in routine care: Ropivacaine 0.375%. A single injection will be performed under ultrasounds. No continuous injection will be performed.
  Interventions: Procedure: distal nerves blocks group; Procedure: Diaphragmatic function assessment

INTERVENTIONS:
Procedure: distal nerves blocks group — * ICB: US probe will be placed just below clavicle inferior to site of needle entry. Following identification of axillary artery and cords, the needle will be advanced posterior to axillary artery. 20 cc of Ropivacaine 0.375% will then be deposited in a U-shaped distribution posterior and to each side of the axillary artery.
  * SSNB will be performed by locating the brachial plexus and the departure of the suprascapular nerve from the superior trunk under the inferior belly of the omohyoid muscle by sliding the transducer distally and then injecting 5 mL of ropivacaine 0.375%.
  * SCNB will be performed injecting 5 mL of ropivacaine 0.375% in the intermuscular plane between the sternocleidomastoid and scalene muscles using a lateral to medial in-plane technique.
Procedure: Diaphragmatic function assessment — Diaphragmatic excursion will be assessed under ultrasound immediately before and after regional anesthesia.
  This a pain free and safe procedure, that we usually perform in patients at risk of respiratory failure.

SUMMARY:
This study aims at assessing the effectiveness of combined suprascapular nerve block (SSNB), infraclavicular brachial plexus block (ICB) and supraclavicular nerve block (SCNB) as surgical anesthesia for patients scheduled for arthroscopic shoulder surgery. The secondary objective is to test the hypothesis that SSNB-ICB-SCNB combination could spare the phrenic nerve.

DETAILED DESCRIPTION:
Material and Methods This study will be performed according to the declaration of Helsinki. The institutional review board of the hospital (Clinique Médipôle Garonne, 45 rue de Gironis, 31036, Toulouse) gave its approval (registration n° 2016-202). Written consent for publication will been obtained from each patient.

Patients This prospective study will be conducted in the Department of Orthopedic surgery of Clinique Médipôle Garonne. Patients will be included from June 2017 to July 2017. Patients undergoing ambulatory arthroscopic shoulder surgery (acromioplasty and supraspinatus tendon repair) will be screened. Exclusion criteria are: age <18 years, brachial plexus neuropathies, acute respiratory distress, coagulopathies, systemic glucocorticoid use, pregnancy, routine use of opioid medications, intolerance for one or more medication of the study protocol and diabetes. All the patients will be operated on by the same surgeon (Dr Duport M.) and regional anesthesia will performed by experienced anesthetists (PM, CC, FF and MM).

Settings Before regional anesthesia (T1), the first sonographic evaluation of the diaphragm will performed.

All patients will be monitored in accordance with current guidelines, including non-invasive blood pressure as well as continuous electrocardiogram and pulse oximetry. The combination of infraclavicular brachial plexus block (ICB) (ropivacaine 0.375%, 20 mL), suprascapular nerve block (SSNB) (ropivacaine 0.375%, 5 mL) and supraclavicular nerve block (SCNB) (ropivacaine 0.375%, 5 mL) will performed. Systemic dexamethasone (10mg) will be administrated in all patients to prolong the analgesic effect of regional anesthesia. Shoulder arthroscopy will be performed in lateral decubitus position. Patients will then be transferred to the post-anesthesia care unit (PACU). Paracetamol (1 g each 6 hours) and Ketoprofen (100mg twice a day) will be systematically administered. Rescue analgesia with tramadol (100mg each 8 hours) will be administered if necessary (verbal rating scale (VRS) >3). Before PACU discharge (T2), a new ultrasonographic diaphragmatic function assessment will be done. Incidence of dyspnea will also be reported.

Patients will be contacted by phone once a day during the first two days after surgery to analyze the time period to the first opioids request, consumption of tramadol tablets and overall satisfaction. Patients will be instructed to keep a diary or write down the time when they took painkillers. Patient satisfaction concerning the procedure will be assessed using an 11-point scale (0: totally unsatisfied, I would definitively want a different anesthesia / analgesia method for the next surgery; 10: totally satisfied, I would definitively want the same anesthesia / analgesia method for the next surgery).

Regional anesthesia procedure Regional anesthesia procedures will be performed with Ultra-Sound (US) equipment (Sonosite Export, Bothell, USA) by experienced anesthetists. The ICB will be performed as follow: after skin disinfection, US probe will be placed just below clavicle inferior to site of needle entry. A 50 mm sonovisible nerve block needle (Ultraplex, B. Braun, Germany) will be inserted using in-plane technique. Following identification of axillary artery and cords, the needle will be advanced posterior to axillary artery. Local anesthetic (LA) (ropivacaine 0.375%, 20 mL) will then be deposited in a U-shaped distribution posterior and to each side of the axillary artery using as few injections as possible.

Then, an in-plane ultrasound-guided SSNB will be performed by locating the brachial plexus and the departure of the suprascapular nerve (SSN) from the superior trunk under the inferior belly of the omohyoid muscle by sliding the transducer distally and then injecting 5 mL of ropivacaine 0.375% in order to surround the nerve with local anesthetic.

As previously described, the SCNB will be performed injecting 5 mL of ropivacaine 0.375% in the intermuscular plane between the sternocleidomastoid and scalene muscles using a lateral to medial in-plane technique. The supraclavicular nerve is a terminal branch of the superficial cervical plexus that supplies the skin overlying the shoulder.

Any instances requiring unscheduled conversion to general anesthesia intraoperatively will be considered as a regional anesthesia failure.

The success of this combination of peripheral nerves blocks is supported by a precise innervation analysis of the shoulder. The anterior aspect of the shoulder joint is supplied by the posterior cord (which provides the subscapular and axillary nerves) and the lateral cord of brachial plexus ( which provides the lateral pectoral nerve). The posterior shoulder joint is innervated by the suprascapular nerve, which originates from the most proximal section of the superior trunk, as well as small branches of the axillary nerve. Combination of ICB and SSNB allows anesthesia of these nerves originating from the brachial plexus. However, cutaneous innervation of the shoulder is complex and partially mediated by the supraclavicular nerve. A block of this terminal branch of the superficial cervical plexus can be easily performed injecting the LA solution in the intermuscular plane between the sternocleidomastoid and scalene muscles.

Ultrasonographic diaphragmatic function assessment Diaphragmatic function will be evaluated using M-mode ultrasonography according to previously described techniques. With the patient in a semi sitting position with the head elevated approximately 30 degrees, diaphragmatic sonography will be performed using a 3.5-5 MHz phased array probe. The probe will be placed immediately below the right or left costal margin in the right or left anterior axillary line and was directed medially, cephalad and dorsally, so that the ultrasound beam reached perpendicularly the posterior third of the corresponding hemi-diaphragm. The two-dimensional (2D) mode will initially be used to obtain the best approach and to select the exploration line; the M-mode will then be used to display the motion of the anatomical structures along the selected line. Patients will be scanned along the long axis of the intercostal spaces, with the liver serving as an acoustic window to the right, and the spleen to the left. Normal inspiratory diaphragmatic movement is caudal, since the diaphragm moves toward the probe; normal expiratory trace is cranial, as the diaphragm moves away from the probe. In M-mode, the diaphragm appeares as a crisp white, hyperechoic line slowly undulating through the respiratory cycle. Patients will be then asked to perform a "voluntary sniff" (VS) test, for which patients will be asked to forcefully inhale through the nose in a sniffing fashion. Diaphragmatic excursion from baseline will be measured in centimeters using the digital calipers on the ultrasound machine interface. A normal upward movement (toward the probe) will be designated positive. A paradoxical downward movement is designated negative. Two measurements will be made, and the largest displacement will be taken as the referred value. The above measurements will be performed immediately preceding nerves blockade, and then just before PACU discharge. As previously described, complete hemi diaphragmatic paralysis is defined as a greater than 75% reduction in diaphragmatic excursion measured in the VS test13. Partial paralysis is defined as a 25% to 75% reduction.

Data analysis Data analysis for this study is largely descriptive, including percentages and counts for categorical data and medians with 25th to 75th interquartile ranges (IQRs) for continuous data. The primary outcome is the success rate of regional anesthesia (i.e. intraoperative conversion to general anesthesia was considered as a regional anesthesia failure). The secondary outcomes are; analysis of diaphragmatic paralysis, dyspnea, post-operative analgesia duration and patient satisfaction. Data were analyzed using Microsoft Excel (Microsoft, Redmond, Washington).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ambulatory arthroscopic shoulder surgery (acromioplasty and supraspinatus tendon repair) will be screened.

Exclusion Criteria:

* Exclusion criteria are: age <18 years, brachial plexus neuropathies, acute respiratory distress, coagulopathies, systemic glucocorticoid use, pregnancy, routine use of opioid medications, intolerance for one or more medication of the study protocol and diabetes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
success of regional anesthesia procedure (no requirement of intraoperative general anethesia) | 12 hours
  The primary outcome is the success rate of regional anesthesia (i.e. intraoperative conversion to general anesthesia was considered as a regional anesthesia failure).
  General anesthesia was defined as requirement of intraoperative invasive ventilation.

SECONDARY OUTCOMES:
diaphragmatic paralysis | 12 hours
  The secondary outcomes is the analysis of diaphragmatic paralysis. Complete hemi diaphragmatic paralysis was defined as a greater than 75% reduction in diaphragmatic excursion measured in the Voluntary Sniff test. Partial paralysis was defined as a 25% to 75% reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Medipole Garonne, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided